CLINICAL TRIAL: NCT00579865
Title: Impact of Biliary Drainage on Quality Of Life in Patients With Malignant Biliary Obstruction
Brief Title: Quality Of Life in Patients With Malignant Biliary Obstruction
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Piera Robson, RN, BSN, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-036
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Gallbladder Cancer; Liver Cancer; Bile Duct Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Gallbladder Neoplasms; Liver Neoplasms; Bile Duct Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group A: Patients scheduled for percutaneous drainage
  Interventions: Behavioral: questionnaires
- Group B: Patients scheduled for a surgical bypass or resection of a high bile duct tumor.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — complete the FACT-Hep, the SSQ, and the Visual Analog Scale for Pruritus Assessment at 1 week and 4 weeks post procedure.
  Groups: Group A
Behavioral: questionnaires — complete the FACT-Hep, the SSQ, and the Visual Analog Scale for Pruritus Assessment at 1 week and 4 weeks post procedure. Patients who have undergone bypass or resection will complete an additional set of questionnaires at 9 and 14 weeks.
  Groups: Group B

SUMMARY:
You may have symptoms like itching, abdominal pain, loss of appetite, fatigue, fevers and chills. The treatment you will receive to relieve the blockage is also intended to relieve symptoms and improve your quality of life. The purpose of this study is to find out if relieving the blockage in your bile duct improves your quality of life.

DETAILED DESCRIPTION:
Malignant biliary obstruction (MBO) may arise in patients with cholangiocarcinoma, pancreatic carcinoma, primary gallbladder carcinoma, hepatocellular carcinoma, or metastatic disease to the liver or portal lymph nodes. MBO is often accompanied by significant symptoms that may result in impairment of health-related quality of life (HRQL), including pruritus, fever, nutritional deficits, abdominal pain, nausea and vomiting, and fatigue. Approaches to the relief of MBO include surgical bypass and/or resection, percutaneous drainage with or without biliary stenting, or endoscopic stenting. The non surgical procedures may be done prior to attempted curative resection or for palliation in individuals with unresectable or recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignant biliary obstruction
* Radiologic or histologic evidence of MBO
* Percutaneous biliary drainage procedure planned or
* Surgical biliary enteric bypass, or hepatic resection with biliary reconstruction (high bile duct tumors) planned
* KPS >50%
* Age 18 years or greater
* Able to speak and read English
* Able to comprehend and execute informed consent
* Prior intervention for MBO not exclusionary

Exclusion Criteria:

* Unable to complete questionnaire due to performance status
* Proxy completion is not accepted
* Medical or psychiatric condition that, in the judgment of the investigator, prevents appropriate comprehension and execution of either the informed consent or the study instrument

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine how surgical or percutaneous drainage affects HRQL scores in patients with MBO, and to determine if these changes are sustained or change over time. | conclusion of the study

SECONDARY OUTCOMES:
To identify factors associated with changes in HRQL after drainage(e.g. diagnosis, level of obstruction, degree of pruritus) | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Piera Robson, RN, BSN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org